CLINICAL TRIAL: NCT05664841
Title: The Impact of a Virtual Magic Trick Training Program on Social Emotional Functioning in Adolescents With Autism
Brief Title: The Impact of a Virtual Magic Trick Training Program
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hon K. Yuen, PhD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1909503-38
Record Dates: First submitted 2022-12-05; First posted 2022-12-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Autism; Pervasive Developmental Disorder
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- magic trick training (Experimental): Participation in a 6 weekly virtual magic trick training camp with three lessons per week.
  Interventions: Behavioral: magic trick training
- waitlist control (No Intervention): Participation in usual daily activities.

INTERVENTIONS:
Behavioral: magic trick training — A typical session will begin with the magician demonstrating a magic trick then revealing the secret move of the trick.The participants will learn and practice each trick. With assistance from the magician, participants will develop an oralstory presentation for the trick. After participants master one trick, the magician will demonstrate and teach the next.
  Arms: magic trick training

SUMMARY:
The proposed project will attempt to confirm the benefits of a structured magic trick training program (MTTP) experience in adolescents with autism. Benefits of participating in a 6-week virtual MTTP will be evaluated using validated assessments to measure social-emotional competencies.

DETAILED DESCRIPTION:
The proposed study will employ a RCT to test the two hypotheses. The design of the MTTP is based on the SEL framework. The study will incorporate a 2 x 3 two-way factorial design with repeated measures at three time points. The two between-subject factor conditions will be participation in a MTTP versus a waitlist control condition that will be evaluated at baseline, immediately post-program, and at 6-week follow-up (within-subject factor conditions). Sixty adolescents with autism will be recruited for this study.

Aim 1. Evaluate the therapeutic benefits of a 6-week virtual MTTP on social-emotional functioning, and emotional stress among adolescents with autism.

Hypothesis #1: Adolescents with autism who participate in a virtual MTTP will demonstrate better social-emotional functioning, and a reduction in emotional stress compared to waitlist controls at the conclusion of a 6-week MTTP.

Hypothesis #2: The positive impact of the virtual MTTP on the participants' improved social-emotional functioning, and reduction in emotional stress will be maintained at 6-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis (with proof of evidence) of autism;
* Aged between 11 and 18 years (younger children may lack the inductive reasoning skills to learn magic tricks);
* Have functional hand dexterity to do magic tricks
* Intact cognition as indicated by a score above the corresponding cut-off point of the child's age on the Mini-Mental Examination for Children; and
* Access to internet and a computer or smartphone that can perform videoconferencing.

Exclusion Criteria:

* Severe hearing or visual impairments that prevent online learning;
* Previous participation in organized magic learning program or camp;
* Current or planned participation in psychological therapy or a clinical trial during the study period that could affect the outcomes of the study.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Test of Adolescents Social Skills Knowledge (TASSK) | baseline
  The TASSK is a self-report 30-item questionnaire that measures knowledge of specific social skills. Scores range between 0 to 26 with higher score reflecting greater knowledge of adolescent social skills.
Test of Adolescents Social Skills Knowledge (TASSK) | at 6 week
  The TASSK is a self-report 30-item questionnaire that measures knowledge of specific social skills. Scores range between 0 to 26 with higher score reflecting greater knowledge of adolescent social skills.
Test of Adolescents Social Skills Knowledge (TASSK) | at 12 week
  The TASSK is a self-report 30-item questionnaire that measures knowledge of specific social skills. Scores range between 0 to 26 with higher score reflecting greater knowledge of adolescent social skills.
Strengths and Difficulties Questionnaire (SDQ) | baseline
  SDQ (peer problem scale and prosocial scale) consists of 10 items rated on a 3-point Likert-type scale (not true=1 to certainly true=3), with higher scores indicating higher psychological problems. Some items require reverse scoring.
Strengths and Difficulties Questionnaire (SDQ) | at 6 week
  SDQ (peer problem scale and prosocial scale) consists of 10 items rated on a 3-point Likert-type scale (not true=1 to certainly true=3), with higher scores indicating higher psychological problems. Some items require reverse scoring.
Strengths and Difficulties Questionnaire (SDQ) | at 12 week
  SDQ (peer problem scale and prosocial scale) consists of 10 items rated on a 3-point Likert-type scale (not true=1 to certainly true=3), with higher scores indicating higher psychological problems. Some items require reverse scoring.
Rosenberg Self Esteem Scale (RSES) | baseline
  RSES consists of 10 items rated on a 4-point Likert-type scale, with higher scores indicate higher self-esteem.
Rosenberg Self Esteem Scale (RSES) | at 6 week
  RSES consists of 10 items rated on a 4-point Likert-type scale, with higher scores indicate higher self-esteem.
Rosenberg Self Esteem Scale (RSES) | at 12 week
  RSES consists of 10 items rated on a 4-point Likert-type scale, with higher scores indicate higher self-esteem.
UCLA Loneliness Scale Version 3 | baseline
  The UCLA Loneliness Scale (Version 3) is a 20-item measure that assesses how often a person feels disconnected from others. Using a 4-point rating scale (1= never; 4 = always), participants answer 20 questions, such as "How often do you feel left out?" and "How often do you feel part of a group of friends?" Researchers later reverse-code the positively worded items so that high values mean more loneliness, and then calculate a score for each respondent by averaging their ratings.
UCLA Loneliness Scale Version 3 | at 6 week
  The UCLA Loneliness Scale (Version 3) is a 20-item measure that assesses how often a person feels disconnected from others. Using a 4-point rating scale (1= never; 4 = always), participants answer 20 questions, such as "How often do you feel left out?" and "How often do you feel part of a group of friends?" Researchers later reverse-code the positively worded items so that high values mean more loneliness, and then calculate a score for each respondent by averaging their ratings.
UCLA Loneliness Scale Version 3 | at 12 week
  The UCLA Loneliness Scale (Version 3) is a 20-item measure that assesses how often a person feels disconnected from others. Using a 4-point rating scale (1= never; 4 = always), participants answer 20 questions, such as "How often do you feel left out?" and "How often do you feel part of a group of friends?" Researchers later reverse-code the positively worded items so that high values mean more loneliness, and then calculate a score for each respondent by averaging their ratings.
Self-efficacy Questionnaire for Children | baseline
  It consists of 16 items rated on a 5-point Likert-type scale (not at all=1 to very well=5) with higher scores indicating higher self-efficacy.
Self-efficacy Questionnaire for Children | at 6 week
  It consists of 16 items rated on a 5-point Likert-type scale (not at all=1 to very well=5) with higher scores indicating higher self-efficacy.
Self-efficacy Questionnaire for Children | at 12 week
  It consists of 16 items rated on a 5-point Likert-type scale (not at all=1 to very well=5) with higher scores indicating higher self-efficacy.
Best Friend Index | baseline
  The Best Friend Index is a scale for the measurement of the features of positive and negative friendship consisting of 18 items. Each item is answered on a 5-point scale (from 1= Never to 5=Very often).
Best Friend Index | at 6 week
  The Best Friend Index is a scale for the measurement of the features of positive and negative friendship consisting of 18 items. Each item is answered on a 5-point scale (from 1= Never to 5=Very often).
Best Friend Index | at 12 week
  The Best Friend Index is a scale for the measurement of the features of positive and negative friendship consisting of 18 items. Each item is answered on a 5-point scale (from 1= Never to 5=Very often).
Quality of Socialization Questionnaire | baseline
  It is a 12-item self-report and parent-report measure to assess the frequency of adolescents get-together, number of friends involved and the level of conflict during get-togethers over the previous month.
Quality of Socialization Questionnaire | at 6 week
  It is a 12-item self-report and parent-report measure to assess the frequency of adolescents get-together, number of friends involved and the level of conflict during get-togethers over the previous month.
Quality of Socialization Questionnaire | at 12 week
  It is a 12-item self-report and parent-report measure to assess the frequency of adolescents get-together, number of friends involved and the level of conflict during get-togethers over the previous month.
Autism Social Skills Profile | baseline
  It is a checklist that provides a comprehensive measure of social functioning of children and adolescents who are on the Autism Spectrum. The 49 items are rated on a 4-point Likert scale with 1=never, 2=sometimes, 3=often, and 4=very often. The test yields three subscale scores: Social/Emotional Reciprocity (SER), Social Participation/Avoidance (SPA), and Detrimental Social Behaviors (DSB), as well as a total score.
Autism Social Skills Profile | at 6 week
  It is a checklist that provides a comprehensive measure of social functioning of children and adolescents who are on the Autism Spectrum. The 49 items are rated on a 4-point Likert scale with 1=never, 2=sometimes, 3=often, and 4=very often. The test yields three subscale scores: Social/Emotional Reciprocity (SER), Social Participation/Avoidance (SPA), and Detrimental Social Behaviors (DSB), as well as a total score.
Autism Social Skills Profile | at 12 week
  It is a checklist that provides a comprehensive measure of social functioning of children and adolescents who are on the Autism Spectrum. The 49 items are rated on a 4-point Likert scale with 1=never, 2=sometimes, 3=often, and 4=very often. The test yields three subscale scores: Social/Emotional Reciprocity (SER), Social Participation/Avoidance (SPA), and Detrimental Social Behaviors (DSB), as well as a total score.
Stanford Social Dimensions Scale | baseline
  The SSDS is more comprehensive, sensitive and specific compared to other instruments in terms of capturing key social processes that are necessary for understanding of social deficits in conditions. The 71 items are rated on a 5-point Likert scale with 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always.
Stanford Social Dimensions Scale | at 6 week
  IThe SSDS is more comprehensive, sensitive and specific compared to other instruments in terms of capturing key social processes that are necessary for understanding of social deficits in conditions. The 71 items are rated on a 5-point Likert scale with 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always.
Stanford Social Dimensions Scale | at 12 week
  The SSDS is more comprehensive, sensitive and specific compared to other instruments in terms of capturing key social processes that are necessary for understanding of social deficits in conditions. The 71 items are rated on a 5-point Likert scale with 1=never, 2=rarely, 3=sometimes, 4=often, and 5=always.

SECONDARY OUTCOMES:
Emotional stress | baseline
  the amount of cortisol in participants' hair.
Emotional stress | at 6 week
  the amount of cortisol in participants' hair.
Emotional stress | at 12 week
  the amount of cortisol in participants' hair.

CONTACTS AND LOCATIONS:
Overall Officials: Hon Yuen, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spencer K, Yuen HK, Jenkins GR, Kirklin K, Vogtle LK, Davis D. The 'magic' of magic camp from the perspective of children with hemiparesis. J Exerc Rehabil. 2021 Feb 23;17(1):15-20. doi: 10.12965/jer.2040802.401. eCollection 2021 Feb. PMID 33728284